CLINICAL TRIAL: NCT03631095
Title: Evaluation of Spinal Metastatic Tumour for Aggressive Spinal Sugery by Dual Energy CT
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805119RINA
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-03

CONDITIONS: Spinal Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Metastatic vertebral disease is a major hazard for oncological patients because the performance and life quality will substantially deteriorate if presence of neoplastic compression. And the subsequent treatment and overall survival will be dismal. Restoration of vertebral stability and prevention of neurological deterioration are treatment goal. Surgical treatment is an important and effective method for metastatic spinal disease. For aggressive surgical method, long-term control is better. However, massive bleeding is often encountered in this surgery, and preoperative evaluation is very important for successful operation. Imaging play major role in this tasks. MRI, angiography, and nuclear medicine studies are common modalities, but take longer time and are often suboptimal. Dual-energy CT has the ability to detect contrast medium enhancement in osseous structure. It therefore is a potential optimal tool in the evaluate the metastatic spinal malignancy. It also own advantage of rapid scanning, optimal resolution, and easy reformatting.In this study, we intend to use this tool to establish the imaging biomarker for tumoural vascularity, to compare its performance with other modalities, and to investigate its optimal imaging condition, which will bring valuable information for treatment planning for aggressive spinal surgery before metastatic disease.

DETAILED DESCRIPTION:
Spinal metastasis is the leading course of vertebral malignancy. It cause neoplastic spinal cord compression and neurological deficit. The treatment strategy depend on the pathological type, performance status, and life expectancy.(1, 2) The goal of treatment is to avoid neurological deterioration, to keep functional life, and to control bone pain. Because disease cure is rarely the treatment goal in the circumstance of metastatic disease, the treatment strategy involve multidisciplinary approaches. When evidence of neoplastic compression, local oncological treatment is often needed to preserve neurological function and to restore vertebral column stability. Radiation therapy can be applied for some radiosensitive tumour, but surgery is often required to meet above goal. Simple decompression and fixation is often applied, but the long-term control rate is suboptimal. Aggressive spinal surgery has relative longstanding effect to maintain neurological and oncological outcome in selective patients. (3)

Aggressive spinal surgery, including extensive corpectomy, vertebrotrectomy, and even spondylectomy, however, is a massive procedure and may result in large amount, sometime life-threatening blood loss. To achieve better surgical outcome and decrease complication, preoperative evaluation needs understanding the detailed skeleton and vascular anatomy. The status of vertebral column stability, extent of tumour involvement, condition of neurological tissue, and vascularity of the tumoural tissue, are all important in determination of the surgical planning and outcome. In many circumstances, preoperative embolization is often required to control blood loss as well.(4, 5) Imaging plays major role in the above information related to the surgical decision and planning.

Current preoperative imaging evaluation include MRI, angiography, bone scan and PET. (6) The MRI is paramount in the spinal imaging. It provides outstanding soft tissue differentiation, which usually depicting the abnormal tumoural tissue clearly. Therefore, MRI stands central role in the surgical evaluation. Nevertheless, in real world, many patients are frail to tolerate lengthy MRI study period, and the MR imaging quality is often suboptimal. For vascular survey, angiography is capable to demonstrate spinal artery and tumour vascularity. Since its relative invasiveness, it is only reserved for patients when preoperative embolization is required or detection of spinal artery is warranted. And because the angiography study for tumour involves selective catheterization of separate segmental artery, the global evaluation of tumoural tissue is not possible. As for nuclear medicine studies, including bone scan and PET, they are highly sensitive and very convenient in detecting multifocal disease. But they are relative non-specific for variable pathology and the spatial resolution is not adequate for surgical evaluation. Therefore, they provide less information when diagnosis has been established.

CT is an important imaging tool for spinal disease. Because of its rapid acquisition, adequate resolution, and easy reformatting, it is optimal for intolerable patients. (7) Nevertheless, osseous structure is extremely radiopaque, evaluation of tumoural enhancement in vertebrae is not easy. It is reserved in special condition, such as detection of vascular structure for embolization and surgery. Recently commercialized dual-energy CT (DECT) can meet the prior result of conventional CT with added value. (8) It uses different energy level simultaneously to image the object. Therefore, optimal bony removal and contrast-noise-ratio can be expected.(9, 10) In spinal disease, it has been used in the detection of marrow edema and compression fracture. (9, 11) On the other hand, material-specific information can be obtained, quantitative evaluation of tumoural enhancement by contrast medium is possible. (12) Along with imaging post-processing technique, DECT can highlight the tumoural part in the background of hyperdense bone. (13) DECT is a promising tool to study the vascularity of the metastatic vertebral tumour. This information is valuable for the surgeon in the decision making and planning for the operation.

We intend to use the dual energy CT in the preoperative evaluation of the vertebral metastasis before aggressive surgery. The research potential and purposes are manifold. First, we want to establish imaging biomarker for tumoural vascularity. Many different enhancement parameters as potential candidate will be measured. Second, we intend to establish one-stop imaging method; therefore, we will compare the diagnostic performance with other imaging modalities. Third, the optimal imaging parameter in the evaluation of bony lesion will be investigated, and many image technical condition will be studied.

Purpose：

1. To establish the quantitative imaging biomarker for vascularity in metastatic vertebral tumour
2. To obtain the optimal DECT scanning parameter and reformatting method in vertebral osseous tumour
3. To provide detailed anatomical information for embolization and surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patient with clinical suspicious for vertebral metastasis and operation is a treatment option
2. Life expectancy more than 6 months
3. Serum creatinine less than 2.0 mg/dL

Exclusion Criteria:

1. Age less than 20 year old
2. Woman in pregnancy or breast feeding
3. Serious allergic reaction to contrast medium

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with vertebral metastasis for aggressive spinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
overall survivial | 5 year
  overall survival after operation

SECONDARY OUTCOMES:
blood loss | one week
  during operation

OTHER OUTCOMES:
local recurrence | 5 years
  local disease after operation

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan